CLINICAL TRIAL: NCT02255253
Title: Efficacy of Telmisartan 40mg and Hydrochlorothiazide 25mg Monotherapy in High Sodium Intake Patients With Mild to Moderate Hypertension: a Multicenter Randomized Double-blinded Parallel Controlled Trial
Brief Title: Telmisartan and Hydrochlorothiazide Antihypertensive Treatment Study in High Sodium Intake Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Puhong Zhang, Associate Professor, The George Institute for Global Health, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013BAI05B02
Record Dates: First submitted 2014-09-24; First posted 2014-10-02 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: Telmisartan; Hydrochlorothiazide; Efficacy; hypertension; high sodium intake
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Long-Term Synaptic Depression; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telmisartan (Experimental): capsule,40mg per day,2 months
  Interventions: Drug: Telmisartan
- Hydrochlorothiazide (Experimental): tablet, 25mg per day, 2 months
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan — capsule,40mg per day,2 months
  Other Names: China Resources Double-crane Pharmaceutical Co., Ltd
  Arms: Telmisartan
Drug: Hydrochlorothiazide — tablet, 25mg per day, 2 months
  Other Names: Tianjin LiSheng Pharmaceutical Co., Ltd
  Arms: Hydrochlorothiazide

SUMMARY:
In this research, the investigators aim to compare the antihypertensive efficacy and safety of monotherapy of routine dose angiotensin receptor antagonist telmisartan (ARB) and diuretic Hydrochlorothiazide (HCTZ) in high sodium intake patients with mild to moderate hypertension. The research will be conducted in the rural area in Hebei province, where people have a high sodium diet in their daily life. The 1200 eligible subjects will be drawn from 12 local county-level hospitals. Subjects will be randomly allocated in double-blind manner into ARB or HCTZ group to be administered telmisartan 40mg per day or hydrochlorothiazide 25mg per day respectively. After two-month treatment, the investigators will evaluate and compare the antihypertensive efficacy and safety between the two therapies.

The first objective of the research is to compare the antihypertensive efficacy of monotherapy of routine dose of angiotensin receptor antagonist telmisartan (ARB) and diuretic Hydrochlorothiazide (HCTZ) in high sodium intake patients with mild to moderate hypertension.The second objective is to compare the safety between the two therapies applied.

Null Hypothesis-H0: There will be no efficacy differences of lowering the systolic pressure between treating high sodium intake patients with mild to moderate hypertension with telmisartan and hydrochlorothiazide.Alternative Hypothesis-H1: There will be efficacy differences of lowering the systolic pressure between treating high sodium intake patients with mild to moderate hypertension with telmisartan and hydrochlorothiazide.

This research is a multicenter randomized double-blinded parallel controlled trial targeting on high sodium intake patients with mild to moderate hypertension in China. The eligible 1200 subjects will be randomly divided into ARB and HCTZ two groups, treated with monotherapy of telmisartan 40mg per day or hydrochlorothiazide 25mg per day respectively. Then, the compliance of the patients will be followed after a week. The investigators will evaluate the efficacy of blood pressure control and the safety of the medicines after one month and two months of the beginning of therapies. Figure 1 shows the research process.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18
* Essential hypertension: systolic blood pressure (SBP) is between 140mmHg-179mmHg and diastolic blood pressure (DBP)<110mmHg OR DBP is between 90mmHg-109mmHg and SBP<180mmHg.
* Hypertension patients diagnosed by spot urine test (urine sodium≥200mmol/24h).
* Subjects are not using antihypertensive medicines or medicines which affect the blood pressure within a week.
* Subjects volunteer to be brought in the research and have signed informed consent form, given that they have understood the research content.

Exclusion Criteria:

* Females who are already pregnant, in lactation and intend to be pregnant.
* Patients who have seriously allergic reaction or angioneurotic edema when taking ARB; Patients who have allergic history of thiazide diuretic (HCTZ) or sulfonamides.
* Patients who do not want to stop or have to take the medicines which are also antihypertensive or affect the blood pressure, other than which provided by the research.
* Stroke or CHD patients who are diagnosed within 6 months. CHD patients are identified by being diagnosed by coronary arteriography or coronary CT angiography, having received coronary stent or coronary artery bypass surgery, or being diagnosed with acute myocardial infarction. Stroke patients are identified by being diagnosed with cerebral thrombosis, cerebral embolism, cerebral hemorrhage, subarachnoid hemorrhage or transient ischemic attack.
* Patients who are clearly diagnosed with following diseases: Congenital disease, myocardiopathy, serious arrhythmia, pulmonary heart disease, various of cardiac failure.
* Patients who are clearly diagnosed with following symptoms or diseases: Proteinuria or heavy proteinuria, renal insufficiency or serious renal function damage, hepatic insufficiency or serious hepatic function damage; retinal exudates or hemorrhage, or papilledema.
* Patients who are clearly diagnosed with serious or deadly diseases in other systems.
* Patients who get dementia or other serious diseases cannot cooperate with researchers.
* Patients who drink 200g white spirits per day in past week.
* Patients who meet other situations which are considered to be inappropriate to be enrolled into the study by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1410 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The difference between 2 groups of the decrease ranges of SBPs before and after the intervention of the subjects | 2 months
  We will measure the SBP for all the participants( around 1400) at baseline and 2\4\8 weeks after intervention with Omron electronic sphygmomanometer HBP - 1300. We will compare the differences between 2 groups at all 4 time points.

SECONDARY OUTCOMES:
The between-group difference of the decrease ranges of DBPs before and after the intervention of the subjects | 2 months
  We will measure the DBP for all the participants( around 1400) at baseline and 2\4\8 weeks after intervention with Omron electronic sphygmomanometer HBP - 1300. We will compare the differences between 2 groups at all 4 time points.

OTHER OUTCOMES:
The between-group difference of the blood pressure control rates before and after the intervention of the subjects | 2 months
  The patients whose SBP is less than 140 (150 for the old) and DBP less than 90 are thought to be controlled.
The between-group difference of the changing ranges of FBG testing results before and after the intervention of the subjects | 2 months
  Blood samples will be collected at baseline and the end of 2-month intervention for FBG test.
The between-group difference of the incidence rates of hypokalemia after the intervention of the subjects | 2 months
  Blood samples will be collected at baseline and the end of 2-month intervention for test

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Pu Hong, Principal Investigator — The George Institute
Locations (14):
- China (14):
  - Chinese Traditional Medicine Hospital of Anguo, Baoding, Hebei
  - Boye hospital, Baoding, Hebei
  - Lixian chinese traditional medicine hospital, Baoding, Hebei
  - Gaoyang hospital, Baoding, Hebei
  - People's hospital in Rongcheng, Baoding, Hebei
  - Mancheng Hospital, Baoding, Hebei
  - Shunping Hospital, Baoding, Hebei
  - People's hospital of Tangxian, Baoding, Hebei
  - Wangdu hospital, Baoding, Hebei
  - Gaobeidian hospital, Baoding, Hebei
  - Central hospital in Baigou, Baoding, Hebei
  - The second hospital of Lai Shui, Baoding, Hebei
  - Wenan Hospital, Lanfang, Hebei
  - Dacheng chinese traditional medicine hospital, Langfang, Hebei

REFERENCES:
- [Derived] Zhang P, Wang H, Sun L, Zhang J, Xi Y, Wu Y, Yan LL, Li X, Sun N. Telmisartan and hydrochlorothiazide antihypertensive treatment in high sodium intake population: a randomized double-blind trial. J Hypertens. 2017 Oct;35(10):2077-2085. doi: 10.1097/HJH.0000000000001407. PMID 28509725